CLINICAL TRIAL: NCT00263055
Title: Multicenter Asia Study in Adjuvant Treatment of Colon Cancer With OxaliplaTin/5FU-LV
Brief Title: MASCOT : Multicenter Asia Study in Adjuvant Treatment of Colon Cancer With OxaliplaTin/5FU-LV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R_9262
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
Safety & tolerability of FOLFOX4 regimen in the adjuvant treatment of colon cancer in Asian patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage Dukes " B2 " (stage II: T3-T4 N0 M0) and " C " (stage III: any T N1-2 M0) colon carcinoma. The inferior pole of the tumor must be above the peritoneal reflection (> 15 cm from the anal margin).
* Patients must have undergone complete resection of the primary tumor without gross or microscopic evidence of residual disease
* Patients must be entered in the study in order to start treatment within 7 weeks after surgery
* Age 18-75 years old
* Performance Status ≤ 2 (Karnofsky > or = 60%)
* No previous chemotherapy, immunotherapy or radiotherapy
* No biological major abnormalities :Absolute neutrophil count > 1.5 x 10^9/l,Platelets ≥ 100 x 10^9/l,Serum creatinine ≤ 1.25 times the upper limit of normal, total bilirubin, ASAT / ALAT < 2 times the upper limit of the normal range,carcinoembryonic antigen < 10 ng/ml.
* Documentation of a negative pregnancy test must be available for premenopausal women with intact reproductive organs
* Men and women who are fertile must use a medically acceptable contraceptive throughout the treatment period and for 3 months following cessation of treatment with oxaliplatin. Subjects must be made aware, before entering this trial of the risk of becoming pregnant or in fathering children
* Signed informed consent obtained prior to study entry

Exclusion criteria

* Pregnant or lactating women
* Women of child bearing potential not using a contraceptive method
* Previous cancer of the colon or rectum
* Previous malignancies other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell carcinoma of the skin, unless there has been a disease-free interval of at least 10 years
* Participation in another clinical trial with any investigational drug within 30 days prior to randomization
* Peripheral neuropathy (NCI CTC [National Cancer Institute Common Toxicity Criteria] > or = Grade I)
* Uncontrolled congestive heart failure or angina pectoris, or hypertension or arrhythmia
* History of significant neurologic or psychiatric disorders
* Active infection

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity | from the inform consent signed up to the end of the study

SECONDARY OUTCOMES:
Occurrence of one or more adverse event in a patient | From the Informed Consent Form (ICF) signature to the end of the study
Overall distribution of intensity of adverse events | from the inform consnet signed up to the end of the study
Occurrence of particular adverse events and their intensities | from the inform consent signed up to the end of the study
Percent of patients completing study treatment | from the inform consent signed up to the end of the study
Percent of patients with grade 1, 2 and 3 neuropathy | at 28 days, 6 months and 12 months after last chemotherapy administration.
Percent of intended dose delivered for 5-FU/LV and Oxaliplatin | from the informed consent signed up to the end of the study
Delays in scheduled dosing | During the study conduct
Dose intensity, as expressed as the amount of 5-FU/LV and Oxaliplatin administered divided by the duration of treatment | during the study conduct
•Survival Analysis •Laboratory assay and vital signs ECOG and KPS | during the study conduct
Long term toxicity | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Claude Valterio, MD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis, Beijing, China
- Sanofi-Aventis, Hong Kong, Hong Kong
- Sanofi-aventis, Seoul, South Korea
- Sanofi-Aventis, Taipei, Taiwan
- Sanofi-Aventis, Bangkok, Thailand